CLINICAL TRIAL: NCT06766526
Title: Internet-based Support for Adjustment to Prostate Cancer (ISAC) - A Randomized Controlled Trial of ICBT for Distress Related to Prostate Cancer
Brief Title: Internet-based Support for Adjustment to Prostate Cancer
Acronym: ISAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Collaborators: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Gerhard Andersson, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISAC
Record Dates: First submitted 2025-01-02; First posted 2025-01-09 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Psychological Distress; Depression - Major Depressive Disorder; Insomnia; Anxiety; Prostate Cancer
Keywords: Psychological distress; Prostate cancer; Cancer; ICBT; Cognitive behavior therapy
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Anxiety Disorders; Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Intervention Model Description: After recruitment finished, participants will be randomized to either tailored ICBT treatment or a control condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tailored ICBT (Experimental): An eight week long ICBT treatment that is tailored to the problem profile of the participant. The treatment is modular, with one module being administered per week of the treatment.
  Interventions: Behavioral: Internet-based cognitive behavioral therapy
- Non-directive support (Active Comparator): The control group will receive weekly support via contact with a therapist, without receiving access to the treatment modules.
  Interventions: Behavioral: Non-directive support

INTERVENTIONS:
Behavioral: Internet-based cognitive behavioral therapy — An eight week ICBT treatment. The treatment is modular and tailored to the problem profile of the participant. One module will be administered every week during the treatment phase.
  Arms: Tailored ICBT
Behavioral: Non-directive support — Participants randomized to this condition will receive weekly support and contact with a therapist via the treatment platform. They will not have access to the treatment modules during the treatment phase.
  Arms: Non-directive support

SUMMARY:
The study aims to study the efficacy of internet-based cognitive behavior therapy (ICBT) in reducing subjective distress and comorbid psychiatric symptoms in men diagnosed with prostate cancer. Participants who have been diagnosed with prostate cancer and are currently not undergoing or scheduled to undergo medical treatment will be recruited. Once recruited, they will be randomized to receive either a tailored, eight-week long ICBT intervention or an attention control group. Both group receive weekly support by a trained therapist.

DETAILED DESCRIPTION:
Men diagnosed with prostate cancer frequently suffer from a wide range of psychological problems that can be traced to their disorder. Examples include depressed mood and worry regarding the prognosis and/or cancer recurrence. Psychological treatments can be used for helping cancer patients deal with this kind of distress, but frequently only targets one kind of symptoms.

This study investigates a tailored approach to providing help for men diagnosed with prostate cancer. Participants randomized to the treatment condition will receive an eight week ICBT intervention which is tailored to the problem profile of the participant in question. The treatment will last eight weeks and participants will receive weekly support and feedback from a therapist. Participants randomized to the control condition will receive weekly therapist support, but not access to the treatment modules. The primary outcome of interest is psychological distress, and other health-related outcomes will be measured as well. Participants will be recruited in Sweden with a nationwide recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Subjectively reported psychological symptoms and problems that have come about after a prostate cancer diagnosis.
* A sum score above 19 on the primary outcome measure (Kessler-10).
* An age of 18 or older.
* Ability to speak, read, and write Swedish.
* Access to a computer/laptop/tablet/smartphone and internet access.
* Sufficient computer profiency to be able to use the treatment platform.

Exclusion Criteria:

* Planned medical treatment or planned change in medication related to the prostate cancer during the treatment period.
* Recently finished (within the past six months) medical treatment for prostate cancer.
* Severe psychiatric or somatic conditions that impedes participation in the study.
* Ongoing substance use problems.
* Acute suicidality.
* Other ongoing psychological treatment.
* Psychopharmaceutic treatment that has been changed within the past month or with planned changes during the treatment phase.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-01-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Kessler-10 (K10) | At pretreatment, weekly during the treatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of psychological distress. Consists of 10 items. Higher scores indicate greater psychological distress. Scores can range between 10 and 50.

SECONDARY OUTCOMES:
Fear of Cancer Recurrence Inventory, short form (FCRI) | At pretreatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of fear of the cancer recurring and/or spreading. Consists of 9 items. Higher scores indicate greater fear/anxiety levels. Scores can range between 0 and 36.
Generalized Anxiety Disorder-7 item scale (GAD-7) | At pretreatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of symptoms of generalized anxiety disorder. Consists of seven items. Higher scores indicate greater anxiety. Scores can range between 0 and 21.
Insomnia Severity Index (ISI) | At pretreatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of insomnia and sleep related-difficulties. Consists of seven items. Higher scores indicate greater sleep related-difficulties. Scores can range from 0 to 28.
Brunnsviken Brief Quality of Life Scale (BBQ) | At pretreatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of quality of life. Consists of 12 items. Higher scores indicate a greater quality of life. Scores can range between 0 and 96.
The EORTC Core Quality of Life questionnaire (EORTC QLQ-C30) | At pretreatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of health-related quality of life. Consists of 30 items and three main subscales which each will serve as an outcome: Global health status, Functional status, and Symptom status. Higher scores indicate a greater health status within the domain. Scores can range between 0 and 100.
The Illness Cognition Questionnaire (ICQ) | At pretreatment, weekly during the treatment, after nine weeks, six months after completion of treatment, and twelve months after completion of treatment.
  Measure of cognitions about the illness (in this case prostate cancer). Consists of 18 items. Analyzed separately as three subscales: Acceptance, Perceived benefits, and Helplessness. Greater scores indicate greater acceptance, more perceived benefits, and greater helplessness, respectively. Will also be used as mediators in a mediation analysis with the rate of change in subscale sum scores used as mediators. Sum scores for each subscale can range between 6 and 24.

OTHER OUTCOMES:
Client Satisfaction Questionnaire-8 item version (CSQ-8) | Measured after nine weeks of treatment.
  Measure of treatment satisfaction. Consists of eight items. Higher scores indicate greater treatment satisfaction. Scores can range between 8 and 32.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Andersson, pHD, Principal Investigator — Linkoeping University
Locations (1):
- Department of Behavioral Sciences and Learning, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Website used for the treatment. — https://www.iterapi.se/sites/isac/